CLINICAL TRIAL: NCT02567981
Title: Impact of the Consumption of an M+ Fortified Premix (Chapuditos®) in 4 Rural Municipalities in the Department of La Libertad, El Salvador in Children From 6 to 59 Months.
Brief Title: Comparison of Two Nutrition Interventions in Young Children in El Salvador
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Mathile Institute for the Advancement of Human Nutrition (Other)
Collaborators: Fundación Salvadoreña para la Salud y el Desarrollo Humano (Other); Humanitas Global Development (Other); Ministry of Health, El Salvador (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-08
Record Dates: First submitted 2015-09-30; First posted 2015-10-05 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Micronutrient Deficiency
Keywords: chronic undernutrition; anemia; micronutrient supplement
MeSH Terms: conditions — Anemia | interventions — ferrous sulfate; Vitamin A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 21 micronutrient fortified supplement (Experimental): 21 micronutrient-fortified supplement
  Interventions: Dietary Supplement: 21 micronutrient-fortified supplement
- Current Standard of Nutritional Care (Active Comparator): Cereal Fortificado (Fortified Cereal) Ferrous sulphate Vitamin A
  Interventions: Dietary Supplement: Cereal Fortificado (Fortified Cereal); Dietary Supplement: Ferrous sulphate; Dietary Supplement: Vitamin A

INTERVENTIONS:
Dietary Supplement: 21 micronutrient-fortified supplement — 21 micronutrient fortified supplement: Dose: 18.75g/day. Contains the following daily amounts per dose: Zinc 9 mg, Copper 300mcg, Iron 12mg, Vitamin D 5 mcg, Folic Acid 160mcg, Vitamin E 5mg, Iodine 90mcg, Calcium 200mg, Vitamin A 250mg, Phosphorus 150 mg, Vitamin C 40mg, Magnesium 40mg, Vitamin B12 0.9mcg, Selenium 17mcg, Thiamine 0.5mg, Manganese 0.17mg, Niacin 6mg, Biotin 8mg, Riboflavin 0.5mg, Vitamin B5 1.8mg, Vitamin B6 0.5 mg. Formula (percentage by weight): Maize 64.08%, Soy Beans 30%, Vitamins and Minerals 5.92%, BHA 0.006%. Energy: 73kcal, Protein 4g, Fat 1g, Dietary Fiber 2g, Carbohydrates 12g.
  Other Names: Chapuditos, M+
  Arms: 21 micronutrient fortified supplement
Dietary Supplement: Cereal Fortificado (Fortified Cereal) — "Cereal Fortificado" Dose: 45g/day. Contains the following daily amounts per dose: Vitamin A 226.6mcg, Thiamine 0.058mg, Riboflavin 0.202mg, Niacin 2.16mg, Panthotenic acid 3.015mg, Vitamin B6 0.765mg, Folate 27mcg, Vitamin B12 0.9mg, Vitamin C 45mg, Vitamin D 1.8mcg, Vitamin E 3.735mg, Vitamin K 45mcg, iron 3.6mg, Zinc 1.8mg, Iodine 18mcg, potassium 180mg, phosphorus 90 mg, calcium 58.50mg. Percentage weight: 58% corn, 20% soy, Skim dry milk 8%, Sugar 9%, Soy Oil 3%, Vitamins and Minerals 0.2%, calcium phosphate 1.23%, Potassium chloride 0.27%. Energy 184.5 kcal, protein 7.2%, Fat 4.1%, Fiber 1.4%, Ash 4.6%.
  Other Names: Cereal Fortificado, Supercereal Plus, FBF-V-10
  Arms: Current Standard of Nutritional Care
Dietary Supplement: Ferrous sulphate — Ferrous sulfate drops children <12 months: 12,5mg elemental iron/day (continuous). Children from 12-23.9months: elemental iron 25mg/day (continuous).
  Chidlren from 24 to 59 months: 1ml/day for two months, every 6 months.
  Arms: Current Standard of Nutritional Care
Dietary Supplement: Vitamin A — Vitamin A Capsules: children <12 months: 100.000 IU/6 months. Children 12-59 months: 200.000 IU/6 months.
  Arms: Current Standard of Nutritional Care

SUMMARY:
Adequate nutrition during the first years of life is essential to reach full body and brain development potential. Children under the age of 5 in Central America and El Salvador suffer from micronutrient deficiencies. In El Salvador, ~ 20% of children under the age of 5 suffer from chronic undernutrition which is reflected in low length-for-their age Z-scores and anemia. This trial will examine the impact on health and growth in young children that will receive either a 21 micronutrient fortified cereal/legume mix manufactured in Guatemala or the current standard of nutritional care. The ultimate goal is to identify other feasible and effective alternatives to prevent micronutrient deficiencies through culturally acceptable vehicles.

DETAILED DESCRIPTION:
A two-arm nutritional intervention trial utilizing a cluster-randomized design will be implemented in the Department of La Libertad, El Salvador, in children from 6 to 59 months of age for 5 years. One arm of the trial will receive a cereal/legume extruded premix fortified with 21 micronutrients (amounts described in Intervention Type section) and the other arm will continue to receive the current standard of nutritional care that consist of a fortified cereal mix, vitamin A capsules, and prophylactic iron drops.

The monitoring and evaluation of this trial will be integrated to an ongoing program implemented by a local NGO (FUSAL) that aims to reduce poverty and micronutrient deficiencies through a variety of strategies. The nutrition products for children under 24 months of age will be provided by El Salvadoran government health workers at the government's health facilities. FUSAL will also be in charge of distributing food products to children from 24 to 59 months of age on a monthly basis at the community sites.

The trial design includes clusters (census subdivisions with a unique number used by the Government of El Salvador to perform the country's census) that were randomized into one of the two treatments. To evaluate the impact of the nutrition interventions, the trial will have two different types of experimental designs:

1. A repeated cross sectional design: to compare outcomes between groups after 1 year and on a yearly basis until the study is completed.
2. Longitudinal design: children will be followed up over time for at least one year, until they turn 60 months and/or the study is completed, to evaluate incidence and recurrence of anemia, undernutrition and morbidity, and other outcomes.

The investigators will test the following hypotheses:

1. Children receiving the 21 micronutrient fortified supplement will have better health and growth than children receiving the nutritional standard of care.
2. Those who receive the 21 micronutrient fortified supplement until 59 months of age continuously will have better health and growth compared to those who received the nutritional standard of care.
3. The effect of the interventions will be most notable in those children who are stunted/anemic.

ELIGIBILITY:
Inclusion Criteria:

* Parental signed informed consent.
* Age 6 to 42 months when study begins (so child can be followed up for at least 1 year).
* Permanent resident of selected municipalities and no intention to move for the next two years.
* Availability and commitment to attend well child visits at government health institutions and to comply to FUSAL's "Libras de Amor" program.

Exclusion Criteria:

* Child has severe wasting (weight for height <-3 z-scores) or any clinical sign/ symptom of severe wasting.
* Child older than 42 months of age when study begins.
* Child has identified conditions that could interfere with their development and growth and/or with severe disease that requires hospital attention.
* Child currently consuming other micronutrient supplements and/or therapeutic foods.
* Child with hemoglobin<7.9g/dL.
* Child participating in another study or program with a nutrition component.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4577 (Actual)
Dates: Start 2015-09; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Changes in mean hemoglobin concentrations | Every six months after enrollment until child reaches 60 months of age or until study completion
Prevalence of anemia | Every six months after enrollment throughout study completion, and/or until child reaches 60 months of age, and/or until study is completed.
  Anemia is defined as hemoglobin <11.0g/dL.
Changes in mean length/height-for age z-scores (HAZ) | Every three months after enrollment throughout study completion, and/or until child reaches 60 months of age.
  Z scores will be calculated based on 2006 child WHO growth standards
Prevalence of stunting defined as HAZ<-2SD below median. | Every three months after enrollment throughout study completion, and/or until child reaches 60 months of age.
  Z scores will be calculated based on 2006 child WHO growth standards
Incidence of acute respiratory tract infections | Monthly from after enrollment throughout study completion, and/or until child reaches 60 months of age.
  Respiratory tract infections definition: any infectious disease of the upper or lower respiratory tract. Caregivers will answer on a monthly basis a brief morbidity questionnaire.
Incidence of diarrhea | Monthly from enrollment throughout study completion, and/or until child reaches 60 months of age.
  Diarrhea definition (WHO): " three or more loose or liquid stools per day (or more frequent passage than is normal for the individual)". Termination of an episode is defined when associated symptoms have been absent for more than 48 hours.
  Caregivers will answer on a monthly basis a brief morbidity questionnaire.

SECONDARY OUTCOMES:
Changes in mean weight-for-height z-scores (WHZ) | Every three months after enrollment throughout study completion, and/or until child reaches 60 months of age.
  Z scores will be calculated based on 2006 child WHO growth standards
Prevalence of wasting defined as (WHZ<-2SD) below the median. | Every three months after enrollment throughout study completion or until child reaches 60 months of age.
  Z scores will be calculated based on 2006 child WHO growth standards
Incidence of wasting defined as (WHZ<-2SD) below the median. | Every three months after enrollment throughout study completion or until child reaches 60 months of age.
  Z scores will be calculated based on 2006 child WHO growth standards
Prevalence of underweight defined as WAZ<-2SD below the median. | Every three months after enrollment throughout study completion or until child reaches 60 months of age.
  Z scores will be calculated based on 2006 child WHO growth standards
Incidence of underweight defined as WAZ<-2SD below the median. | Every three months after enrollment throughout study completion or until child reaches 60 months of age.
  Z scores will be calculated based on 2006 child WHO growth standards
Changes in mean WAZ | Every three months after enrollment throughout study completion, and/or until child reaches 60 months of age.
  Z scores will be calculated based on 2006 child WHO growth standards
Prevalence of overweigth defined as BMI-for-age z score>2SD above median. | Every three months after enrollment throughout study completion or until child reaches 60 months of age.
  Z scores will be calculated based on 2006 child WHO growth standards
Incidence of overweigth defined as BMI-for-age z score>2SD above median. | Every three months after enrollment throughout study completion or until child reaches 60 months of age.
  Z scores will be calculated based on 2006 child WHO growth standards
Changes in mean BMI-for-age z score | Every three months after enrollment throughout study completion or until child reaches 60 months of age.
  Z scores will be calculated based on 2006 child WHO growth standards
Length/Height gain/month (cms) | Every three months after enrollment throughout study completion or until child reaches 60 months of age.
Weight gain/month (Kg) | Every three months after enrollment throughout study completion or until child reaches 60 months of age.
  Z scores will be calculated based on 2006 child WHO growth standards
Prevalence of respiratory tract infections and of diarrhea | Monthly after enrollment throughout study completion or until child reaches 60 months of age.
  Caregivers will answer on a monthly basis a brief morbidity questionnaire. Data from health cards will also be recorded.
Incidence of Stunting (HAZ<-2SD) | Every three months after enrollment throughout study completion or until child reaches 60 months of age.

OTHER OUTCOMES:
Caregiver's practices related to infant and young child feeding, hygiene and sanitation | Baseline- 6 months - 12 months - 18 months - 24 months from enrollment.
  In a subsample of randomly selected participants infant/child feeding practices will be measured through home observation visits and semi-structured questionnaires.
Milestone development score differences assessed through a developmental milestone scale | Every 6 months after enrollment throughout study completion or until child reaches 60 months of age.
  A milestone developmental scale that has been adapted to the local context will be implemented every 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Reinhart, PhD, Principal Investigator — The Mathile Institute for the Advancement of Human Nutrition
Locations (1):
- FUSAL, Santa Elena, El Salvador